CLINICAL TRIAL: NCT02451761
Title: Molecular Characterization of Apparently Balanced Chromosomal Rearrangements by Next-generation Sequencing in 55 Patients With Intellectual Disability and/or Multiple Congenital Anomalies
Brief Title: Apparently Balanced Chromosomal Translocation/ Next-generation Sequencing/ Intellectual Disability
Acronym: ANI
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 2014.858
Record Dates: First submitted 2015-05-06; First posted 2015-05-22 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2016-08

CONDITIONS: Intellectual Disability; Congenital Abnormalities
Keywords: chromosomal rearrangement; next generation sequencing; intellectual disability; multiple congenital anomalies; gene disruption
MeSH Terms: conditions — Intellectual Disability; Congenital Abnormalities; Abnormalities, Multiple | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sequencing: Blood sampling will be carried out in all patients ; molecular analysis and sequencing will be performed on these samples
  Interventions: Biological: Blood sampling

INTERVENTIONS:
Biological: Blood sampling

SUMMARY:
Apparently balanced chromosomal rearrangement (ABCR) associated with an abnormal phenotype is a rare but problematic event. It occurs in 6% of de novo reciprocal translocations and 9% of de novo inversions. Abnormal phenotype, including intellectual disability and / or multiple congenital anomalies (ID/MCA) may be explained either by associated cryptic genomic imbalances detectable by array-CGH or by gene disruption at the breakpoint. However, breakpoint cloning using conventional methods (i.e., fluorescent in situ hybridization (FISH), Southern blot) is often laborious and time consuming and cannot be performed routinely. Without complete investigation of these rearrangements, genetic counseling is a real challenge. Recently, the investigators and others showed that Next-Generation Sequencing (NGS) is a powerful and rapid technique to characterize ABCR breakpoints at the molecular level.

The ANI project (ABCR NGS ID) aims at characterizing at the molecular level ABCR in 55 patients presenting with intellectual disability and/or multiple congenital anomalies (ID/MCA) using NGS. The investigators make the hypothesis that ABCR account for the patient phenotype, either by gene disruption or position effect, since genomic imbalance would have been previously excluded by array-Comparative Genomic Hybridization (CGH).

The ANI project is a 3-year-long study that will be conducted by a consortium of 21 partners, including 19 french hospital cytogenetics laboratories, a research team (TIGER), and a cellular biotechnology center. Patients will be recruited by each Cytogenetics laboratory. ABCR breakpoints will be molecularly characterized by NGS and a first bio-informatics analysis. The results will be verified by amplification of junction fragments by polymerase Chain Reaction (PCR) followed by Sanger sequencing, allowing the localization of breakpoints at the base-pair level. In some complex cases, FISH experiment will be necessary to clarify the results. A second bio-informatics analysis will then determine breakpoints' characteristics (sequence, repeated elements, gene and regulatory elements). Finally, for each breakpoint, gene expression studies will be performed including the gene disrupted by the breakpoint and two neighboring genes. All these data, together with those already available in the literature and databases will be integrated to determine if the gene could account for the patient's phenotype, allowing an appropriate genetic counseling.

This project will identify new candidate genes involved in ID and developmental anomalies. It will also contribute to the development and evaluation of NGS as a diagnostic tool for ABCR and ID/MCA. It will also allow unraveling mechanisms and functional consequences of ABCR, in particular in term of position effect.

In conclusion, the ANI project will contribute to the improvement of diagnostic management and genetic counseling of patients with ID/MCA and ABCR. It will also contribute to the understanding of ABCR physiopathology and to the unraveling of pathway involved in development and brain function, thus improving genetic counseling for ID/MCA patients in general.

ELIGIBILITY:
Inclusion Criteria:

* Abnormal phenotype: intellectual disability and/or multiple congenital anomalies.
* Post-natal cases
* ABCR diagnosed by standard karyotype, including reciprocal translocation, inversion, insertion and Complex Chromosomal Rearrangement (CCR).
* de novo ABCR. Inherited ABCR could be included if the transmitting parent shows also an abnormal phenotype or if the rearrangement involves an imprinted chromosome.
* Array-CGH results normal that mean absence of pathogenic imbalances. Identification of Variant Of Unknown Significance (VOUS) does not prevent from inclusion.
* Information and written consent of patient or his legal representative (information and consent form available on request).
* Covered by a Health System

Exclusion Criteria:

* Pathogenic genomic imbalance demonstrated by array-CGH.
* Identification of an independent etiology (i.e. monogenic disease, environment,…).
* Rejection to participate ton the study
* Weight inferior to 6 kg

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting intellectual disability and/or multiple congenital anomalies
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2015-04; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Identification of candidate genes and genes responsible for the phenotype disrupted at the breakpoints | At the end of the study (36 months)
  Blood samples will be collected at inclusion ; analysis wil be performed at the end of the study (between 30 and 36 months)

SECONDARY OUTCOMES:
Development of a routine bio-informatic protocol for analysis of ABCR by NGS | At the end of the study (36 months)
  Ratio between the number of breakpoints detected by both karyotype ans NGS and the number of breakpoints detected by karyotype alone.
Number of patients presenting at least one disrupted gene | At the end of the study (36 months)
  This outcome will help us ti confirm the NGS performance for the detection of breakpoints of ABCR.
Number of patients for which a diagnosis could be performed | At the end of the study (36 months)
  Number of patients for which a diagnosis could be performed (responsible gene) compared to the total number of patients. This ration will be compared to a reference raio of 10% by a unilateral test. This will allow us to evaluate a next-generation sequencing strategy in clinical context (diagnostic yield)

CONTACTS AND LOCATIONS:
Locations (1):
- laboratoire de Cytogénétique Constitutionnelle - Centre de Biologie et Pathologie Est, Bron, France

REFERENCES:
- See also: Related Info — http://www.agence-nationale-recherche.fr